CLINICAL TRIAL: NCT05850026
Title: Mitral Regurgitation in Hypertrophic Obstructive Cardiomyopathy: Fix it in a Simple, Effective and Durable Way!
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: MIHOC
Record Dates: First submitted 2023-01-27; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy; Mitral Regurgitation
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Septal myectomy and mitral valve repair with edge-to-edge technique — Resection of the obstructing part of the interventricular septum and mitral repair using the edge-to-edge technique (suture of leaflets free margins in the regurgitation spot)

SUMMARY:
Septal myectomy is performed in selected cases to treat patients with hypertrophic obstructive cardiomyopathy (HOCM). The mechanism that causes obstruction involves both the outflow tract itself and the mitral apparatus, with the appearance of mitral regurgitation (MR) by SAM (Systolic Anterior Motion).

When the interventricular septum is not particularly thick, isolated myectomy may not be sufficient to eliminate the SAM; in these cases the concomitant treatment of the mitral valve is considered. Different approaches have been proposed: mitral replacement with prosthesis, plication or lengthening of the anterior leaflet or the edge-to-edge (EE) technique.

In addition, a small proportion of patients with HOCM may have MR from organic valve abnormalities, requiring specific treatment.

Currently, there are few studies in the literature aimed at determining the role of EE in the context of HOCM; most of these studies are characterized by short follow-up or by the scarcity of echocardiographic data.

The aim of the present study is to evaluate the long-term outcomes of EE associated with septal myectomy in patients with CMIO, both from a clinical point of view and by reporting echocardiographic data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HOCM with indication for surgery,
* patients operated on from 2000 to 2017
* contextual diagnosis of MR needing reparative surgical treatment
* age ≥ 18 years

Exclusion Criteria:

* hypertophic left ventricle due to other causes (aortic stenosis, arterial hypertension)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with HOCM and MR, who underwent concomitant septal myectomy and mitral valve repair with edge-to-edge technique
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Survival time after intervention | through study completion, a minimum of 2 years
freedom from reintervention | through study completion, a minimum of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No